CLINICAL TRIAL: NCT05128552
Title: Effect of Lung Volume Recruitment Technique on Cough Efficacy in Postextubated Patients With Ineffective Cough
Brief Title: Effect of Lung Volume Recruitment Technique After Extubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud El-Sayed Abduh Ragab, ICU Physical Therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LVR in ICU
Record Dates: First submitted 2021-10-29; First posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Mechanical Ventilation Complication; Diaphragm Issues; Cough; Ineffective Airway Clearance; Intensive Care Unit Acquired Weakness
Keywords: Cough peak flow; Lung volume recruitment; Air stacking; Cough efficacy; Post extubated patient; Respiratory therapy; Intensive care unit; Mechanical ventilation
MeSH Terms: conditions — Cough

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Twenty-five patients who received traditional chest physiotherapy and LVR technique for 30-45 minutes for successive 4 Days after extubation
  Interventions: Device: Lung volume recruitment technique; Other: Traditional chest physiotherapy
- Control group (Active Comparator): Twenty-five patients who received only traditional chest physiotherapy for 30 minutes at least for successive 4 Days after extubation
  Interventions: Other: Traditional chest physiotherapy

INTERVENTIONS:
Device: Lung volume recruitment technique — A self inflating Ambu bag with one way valve , augmentation volume of air within 3 to 4 successive breaths and holding few seconds then coughing
  Other Names: Air stacking or breath stacking technique
  Arms: Study group
Other: Traditional chest physiotherapy — Positioning of the patient according the drainage position for each lobe of each lung and applying airway hygiene techniques such as percussion and vibration

SUMMARY:
This study was conducted to investigate the effect of the LVR technique on cough ineffectiveness, to determine its benefit as a simple, safe, and inexpensive cough augmentation technique, and to determine how much the LVR method, for augmenting CPF, is useful in enhancing the success of extubation and reducing the rate of reintubation.

DETAILED DESCRIPTION:
An effective cough is so vital in protecting against respiratory tract infections, so the importance of an intact cough mechanism is reflected in the occurrence of pulmonary problems which are the most common cause of hospital admission in people with respiratory muscle weakness who are unable to cough effectively. Ineffective cough results in a tendency to retain bronchial secretions and an increased risk of pulmonary complications, such as frequent or recurrent pneumonia, atelectasis, and infectious respiratory problems.

Cough flow testing (expiratory flows testing) is useful as a monitoring or diagnostic tool in clinical practice and research. Both peak expiratory flows (PEF) and cough peak flows (CPF) have been described as useful clinical measures of respiratory muscle function and cough effectiveness. Cough peak flow (CPF) gives an important measure of the cough strength which determines the effectiveness of cough. It is the maximum expiratory flow recorded immediately following the opening of the glottis during normal cough. Cough effectiveness is suboptimal when cough peak flow (CPF) is less than 270 L/min.

Mechanical Ventilation "MV" has deleterious effects caused by the endotracheal intubation, including changes in mucociliary clearance and inhibition of the coughing mechanism which, in turn, favor areas of hypoventilation and atelectasis, thus increasing the risk of ventilator-associated pneumonia. Respiratory compromise due to recurrent atelectasis, inability to clear secretions, and respiratory infections also increase morbidity and mortality. Prolonged MV results in respiratory muscle dysfunction shown in diaphragmatic atrophy and contractile dysfunction (ic., Ventilator-induced diaphragmatic dysfunction "VIDD") affecting the ability of the person to cough effectively. Indeed, the onset of VIDD in both animals and humans is rapid as significant diaphragmatic atrophy and contractile dysfunction occur within the first 24 - 48 h of MV. Although suctioning of secretions from the trachea to remove tracheobronchial and upper airway secretions is the standard of care, this method is ineffective for clearing peripheral airways and basal retained secretions.

The clinical practice guides referred to patients with respiratory muscles weakness like after prolonged MV and in neuromuscular diseases recommend the usage of cough augmentation and mucociliary clearance techniques in patients with CPF < 4.5 L/s (270 L'min) and using such techniques continuously in patients with CPF < 2.7 L/s (160 L/min). Cough augmentation techniques such as LVR are supposed to be used to reinforce cough effectiveness, particularly for patients with prolonged mechanical ventilation. So, the importance and strength of this study are to assess the effects of the LVR technique as a cough augmentation mean on CPF of post-extubated patients with an ineffective cough which can cause risky respiratory complications may lead to death in confronting to effects of traditional chest physiotherapy and suctioning and therefore, their therapy or management program can be precisely and appropriately planned. Moreover, the identification of effective, safe measures to optimize cough efficacy is, therefore, key to improving quality of life and minimizing morbidity & mortality rates in those patients. Additionally, as a secondary purpose to determine how much the LVR method, for augmenting CPF. is useful in enhancing the success of extubation and reducing the rate of re-intubation that indicated if extubation failure occurred.

ELIGIBILITY:
Inclusion Criteria:

* Forty to sixty years old patients had undergone mechanical ventilation for ≥ 48 hours in a controlled mode and had been weaned after a successful spontaneous breathing trial with suboptimal or poor CPF < 270 L/min.
* Patients were able to assume a sitting position.
* All participants were aware, cooperative, competent, able to comply with treatment, and able to understand and follow instructions.

Exclusion Criteria:

* Presence of significant or active hemoptysis, untreated or recent pneumothorax, bullous emphysema, lung trauma, or recent lobectomy.
* Patients with comorbidities interfering and compromising the success of either weaning or extubation, like cardiac arrhythmia, pericardial effusion, congestive heart failure, or acute coronary syndrome.
* Patients who had originally inadequate training performance of the respiratory muscle such as those having NMD, i.e., myopathy or neuropathy.
* Impaired consciousness/inability to communicate.
* Patients who had a neurological deficit resulted in bulbar affection.
* Patients with indications for MV, but contraindicated for physical therapy like pulmonary embolism.
* Patients who had undergone tracheotomy before extubation also were excluded or who had experienced less than 24 hours of mechanical ventilation.
* Patients with unstable hemodynamics or cardiac instability.
* Current undrained pleural effusion or previous pneumothorax or barotrauma.
* Uncontrolled severe COPD, poorly controlled asthma, and severe bronchospasm.
* Patients with visual or/and auditory problems.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Cough peak flow rate | "Day 4"
  The maximum expiratory flow produced immediately after the glottis opens during a physiological cough
Peak expiratory flow rate | "Day 4"
  The maximum rate at which the air can be expired after a deep inspiration
Oxygen Saturation | "Day 4"
  The percentage that represents how haemoglobin are saturated with oxygen atoms

SECONDARY OUTCOMES:
Extubation's success | "Day 4"
  The patient pass first 48 - 72 hours after extubation alive and doesn't need to be reintubated

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud S. Ragab, Bsc, Principal Investigator — Cairo University
Locations (1):
- Faculty of physical therapy Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rose L, Adhikari NK, Leasa D, Fergusson DA, McKim D. Cough augmentation techniques for extubation or weaning critically ill patients from mechanical ventilation. Cochrane Database Syst Rev. 2017 Jan 11;1(1):CD011833. doi: 10.1002/14651858.CD011833.pub2. PMID 28075489
- [Background] Rose L, Adhikari NK, Poon J, Leasa D, McKim DA; CANuVENT Group. Cough Augmentation Techniques in the Critically Ill: A Canadian National Survey. Respir Care. 2016 Oct;61(10):1360-8. doi: 10.4187/respcare.04775. Epub 2016 Sep 13. PMID 27624630